CLINICAL TRIAL: NCT04339959
Title: Remote Assessment of Physical Function in Older Cancer Survivors
Brief Title: Remote Assessment of Physical Function
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UNM HSC IRB 17-334; K07CA215937-02 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cancer Survivors
Keywords: physical function; physical performance; video conferencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phase I: First, we will test proof-of-concept that participants will be able to follow the testing protocol and use the tablet computer to communicate with the investigator (10-12 participants). The test protocol will be refined based on what is learned after a minimum of 10 participants. We anticipate no more than 12 participants needed for this phase.
  Interventions: Other: Remote Assessment of Physical Function with Direct Observation
- Phase II: Next, 10-20 new participants will be enrolled to evaluate the validity of videoconference vs. face-to-face assessment (i.e., direct observation) of physical performance. Communication will occur between the remote assessor and the participant. The direct observer will not communicate directly to the participant, unless there is a safety issue. After completing 10 participants without a major change in the test protocol, we will proceed to the next phase.
  Interventions: Other: Remote Assessment of Physical Function with Direct Observation
- Phase III: This phase involves participants repeating the test protocol, but without the face-to-face assessment (i.e., direct observation). This will test the ability of the participant to receive the box of test instructions and materials in the mail, unpack the box, communicate with the remote assessor via videoconferencing, pack up the box, and return it (postage paid) to the study team. This step will involve 5-10 participants from Phases 1 and 2, who have provided approval for future contact (see approved Future Contact form). Once 5 participants have successfully and safely completed the test protocol, we will proceed to Phase 4.
  Interventions: Other: Remote Assessment of Physical Function
- Phase IV: This phase is the same as Phase 3, except it includes newly enrolled participants, i.e., representing the first-time participants have enrolled/participated in this study. This will eliminate the practice effect that will occur in phase 3. This step will enroll 5-10 participants.
  Interventions: Other: Remote Assessment of Physical Function

INTERVENTIONS:
Other: Remote Assessment of Physical Function with Direct Observation — An android tablet with Wi-Fi and cellular will be used to compare videoconferencing with face-to-face assessment of 2 timed, physical performance tests. The physical performance tests include the 30-second chair stand test (30s-CST) and the Timed Up & Go (TUG) test. The TUG test is measured as the time to stand from a standard arm chair, walk 10 feet, turn around, return to start and sit down. The 30s-CST is measured as the number of times a person comes to a full standing position from a chair in 30 seconds, as quickly as possible, without using ones' hands.
  Groups: Phase I; Phase II
Other: Remote Assessment of Physical Function — An android tablet with Wi-Fi and cellular will be mailed to study participants to remotely assess 2 timed, physical performance tests. The physical performance tests include the 30-second chair stand test (30s-CST) and the Timed Up & Go (TUG) test. The TUG test is measured as the time to stand from a standard arm chair, walk 10 feet, turn around, return to start and sit down. The 30s-CST is measured as the number of times a person comes to a full standing position from a chair in 30 seconds, as quickly as possible, without using ones' hands.
  Groups: Phase III; Phase IV

SUMMARY:
The primary objective is to evaluate the validity and reliability of using videoconferencing to assess physical performance tests self-administered by older cancer survivors in their own homes. This remote assessment will be compared to the traditional face-to-face (i.e., in-person) assessment and to accelerometer data.

DETAILED DESCRIPTION:
The ultimate goal of this research study is to develop a test protocol to allow older cancer survivors to self-administer physical performance tests in the survivor's own home, while an investigator remotely assesses the tests via videoconferencing. The test protocol includes written and video instructions and the test kit. To achieve this objective, the study will proceed with a series of phases. A similar concept of "saturation" will be applied, as is done in qualitative studies. In qualitative studies, the number of focus groups or interviews is based on the saturation point, i.e., the point at which no new information is learned. For the current study, each study phase will include a range in the number of participants enrolled. At the point at which no new information is being learned, i.e., no further adjustments are needed to the test protocol, the study will proceed to the next phase.

ELIGIBILITY:
Inclusion Criteria:

* Residence in New Mexico
* Previous diagnosis of cancer, completed primary treatment (surgery, radiation, chemotherapy), and not currently being treated for a recurrence.
* Mild-to-moderate physical functional impairment (≥2 functions limited a lot or limited a little on the Short Form 36-item Physical Function Subscale)
* Able to speak, read, & understand English
* Participating in less than 120 minutes per week of moderate-to-vigorous intensity physical activity
* Living independently and capable of walking 3 blocks without stopping to rest.
* Availability of a family member or friend to be present (for safety) during remote assessment of performance tests (Phases III and IV only)
* No severe impairments or pre-existing medical limitations for engaging in daily light-intensity physical activity (e.g., severe orthopedic conditions, pending hip/knee replacement, chronic vertigo, dementia)
* No severe hearing or vision deficits that would inhibit communication with the research team via videoconferencing and tablet use.
* Willing to use a tablet computer and videoconferencing software to communicate with a study team member during the assessment.
* Enough space (14 feet by 3 feet) to safely conduct the physical function tests.
* Not at high risk for falls

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-11-13 (Actual); Study Completion 2021-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy K Blair, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blair CK, Harding E, Herman C, Boyce T, Demark-Wahnefried W, Davis S, Kinney AY, Pankratz VS. Remote Assessment of Functional Mobility and Strength in Older Cancer Survivors: Protocol for a Validity and Reliability Study. JMIR Res Protoc. 2020 Sep 1;9(9):e20834. doi: 10.2196/20834. PMID 32769075

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase III: This phase involves participants repeating the test protocol, but without the face-to-face assessment (i.e., direct observation). A sample of participants from earlier phases were enrolled/consented (a second time) to participate in Phase III. This will test the ability of the participant to receive the box of test instructions and materials in the mail, unpack the box, communicate with the remote assessor via videoconferencing, pack up the box, and return it (postage paid) to the study team. This step will involve 5-10 participants from Phases 1 and 2, who have provided approval for future contact (see approved Future Contact form). Once 5 participants have successfully and safely completed the test protocol, we will proceed to Phase 4.
  Remote Assessment of Physical Function: An android tablet with Wi-Fi and cellular will be mailed to study participants to remotely assess 2 timed, physical performance tests. The physical performance tests include the 30-second chair stand test (30s-CST) and the Timed Up & Go (TUG) test. The TUG test is measured as the time to stand from a standard arm chair, walk 10 feet, turn around, return to start and sit down. The 30s-CST is measured as the number of times a person comes to a full standing position from a chair in 30 seconds, as quickly as possible, without using ones' hands.
Period: Overall Study
Arm/Group | Phase I | Phase II | Phase III | Phase IV
Started | 10 | 5 | 9 | 9
Completed | 10 | 5 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Phase III | Phase IV | Total
Number analyzed (Participants) | 10 | 5 | 9 | 9 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 0 | 1 | 3
  >=65 years | 8 | 5 | 9 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 7 | 6 | 22
  Male | 3 | 3 | 2 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race-Ethnicity: non-Hispanic White | 10 | 4 | 9 | 8 | 31
  Race-Ethnicity: Hispanic White | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 9 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Validation - 30-second Chair Stand Test
Description: Comparison of remote assessment to the traditional face-to-face (i.e., in-person; direct observer) assessment. Phase 2 will enroll 10-20 participants, depending on the point at which no new information is learned about the use of the toolkit (including instructions). Comparisons will be made between the direct observer and the remote assessor. The 30-second chair stand test involves standing up from a chair and sitting down as quickly and safely as possible, preferably without the use of upper extremity support. It is measured by the number of times a person comes to a full standing position from a chair in 30 seconds. The outcome is the difference in the number of chair stands counted between the direct observer and the remote assessor.
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: chair stands
Groups:
- Phases I and II: Combined proof of concept and validation phases since the validation phase was stopped in March of 2020 due to the COVID-19 pandemic.
Arm/Group | Phases I and II
Number analyzed (Participants) | 15
chair stands | 0.33 [-1.56 to 0.9]

2. Primary Outcome: Validation - Timed Up & Go Test
Description: Comparison of remote assessment to the traditional face-to-face (i.e., in-person; direct observer) assessment. Phase 2 will enroll 10-20 participants, depending on the point at which no new information is learned about the use of the toolkit (including instructions). The Timed Up & Go test involves standing up from a standard armchair, walking 10 feet, turning around (180° turn), and walking back to the chair and sitting down. Comparisons will be made between the direct observer and the remote assessor. The outcome is the difference in the number of seconds counted between the direct observer and the remote assessor.
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Phases I and II
Number analyzed (Participants) | 15
seconds | 1.27 [0.28 to 2.26]

3. Secondary Outcome: Reliability - Percentage of Participants Who Successfully Completed the Revised Protocol.
Description: Test of whether a sample of participants from Phases I & II can repeat the test protocol 2-3 months later. This phase will enroll 5-10 participants. The outcome is subjective -- whether the participant could successfully receive the test kit, follow the instructions, communicate with the remote assessor, and perform the two measure of physical performance.
Time Frame: 3 months
Population: Phase III is the test of reliability, i.e., whether a select number of participants from the earlier phases can repeat the revised test protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I | Phase II | Phase III | Phase IV
Number analyzed (Participants) | 0 | 0 | 9 | 0
Participants |  |  | 9 |

ADVERSE EVENTS:
Time Frame: Through study completion (from date of receipt of study toolkit until completion of assessment; up to 1 week)
Arm/Group | Phase I | Phase II | Phase III | Phase IV
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT04339959/Prot_SAP_000.pdf